CLINICAL TRIAL: NCT01051791
Title: Phase II Study of RAD001 for Treatment of Refractory, Recurrent, Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Phase II Study of RAD001 Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Julie E. Bauman, MD, MPH (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Julie E. Bauman, MD, MPH, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-032
Record Dates: First submitted 2010-01-18; First posted 2010-01-20 (Estimated); Results first posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-11

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: RAD001; Everolimus
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus 10 mg daily (Experimental): The study of the efficacy of everolimus will proceed in two stages after the method of Simon1. In the first stage 15 patients will be accrued and treated. If 9 or fewer patients show clinical benefit the study will be terminated. If 10 or more patients show clinical benefit the study will proceed to the second stage, accruing an additional 26 patients. If the second stage is complete and a total of 29 or more patients show clinical benefit among the 41 patients treated, the treatment CBR for will be considered high enough to warrant further study. Conversely, if the evaluation of everolimus concludes at the first stage, or if 28 or fewer patients experience a clinical benefit after completing the second stage, the therapy will not be considered for further study.
  1
  Interventions: Drug: Everolimus 10mg daily

INTERVENTIONS:
Drug: Everolimus 10mg daily — RAD001 is a pill that will be taken orally (by mouth), at a dose of 10 mg, once a day for 28 days.
  Other Names: Everolimus

SUMMARY:
To carry out exploratory studies to determine if activity of this regimen correlates with tumor and patient associated markers of the EGF-R/mTOR pathway These markers may correlate with activity of this regimen and provide exploratory insights in to the mechanism of this treatment approach.

Expression of the pathway components including EGF-R and phosphorylated EGF-R (p-EGF-R), ERK and p-ERK, Akt and p-Akt(T308 and S473), p70s6k and p-p70s6k, S6 and p-S6, HIF-1-alpha, p27 and 4E-BP1 will be assessed. Mutation and FISH analysis for EGF-R expression will also be performed on tumor samples. Biopsies will be obtained at the following times: pre-treatment, and after 4 weeks (one cycle) of treatment. If available, original diagnostic tissue may be submitted in place of the pre-treatment biopsy.

DETAILED DESCRIPTION:
The study of the efficacy of RAD001 will proceed in two stages after the method of Simon . In the first stage 15 patients will be accrued and treated. If 9 or fewer patients show clinical benefit the study will be terminated. If 10 or more patients show clinical benefit the study will proceed to the second stage, accruing an additional 26 patients. If the second stage is complete and a total of 29 or more patients show clinical benefit among the 41 patients treated, the treatment CBR for will be considered high enough to warrant further study. Conversely, if the evaluation of RAD001 concludes at the first stage, or if 28 or fewer patients experience a clinical benefit after completing the second stage, the therapy will not be considered for further study.

Current knowledge about the molecular mechanisms of cancer-related pathways involved in cellular signaling, cell cycle regulation and cell death is yielding therapies directed at specific components of these pathways, such as the epidermal growth factor receptor (EGF-R), the mammalian target of rapamycin (mTOR), the vascular endothelial growth factor receptor (VEGF-R) and the insulin-like growth factor receptor (IFG-R). Both small molecule and monoclonal antibody therapies directed against these targets are available. Furthermore, immunohistochemistry (IHC), fluorescence in situ hybridization (FISH) and mutation analysis are available for profiling expression of pathway components, raising the possibility of individualized prognosis and therapy.

One receptor in particular, is both a prognostic factor and a therapeutic target in HNSCC. Upregulation of EGF-R expression and aberrant activation of kinase cascades downstream of this receptor occur early in the process of carcinogenesis and play a major role in malignant progression.1 The level of EGF-R expression correlates with recurrence and poor prognosis in HNSCC. A well tolerated anti-EGF-R monoclonal antibody, cetuximab, has shown remarkable activity against HNSCC, including statistically significant improvement in survival for patients with locally advanced disease treated with radiotherapy, leading to its regulatory approval for this disease.2 Unfortunately, despite survival advances achieved with EGF-R inhibitors, the majority (~60%) of patients with advanced disease are refractory to EGF-R directed therapies.3 One anticipated mechanism by which the current regimen may fail in some patients is the upregulation of escape pathways downstream of the EGF-R. A pathway of particular interest is the PI3/AKT/mTOR axis, within which the mTOR protein may be targeted by the tyrosine kinase inhibitor RAD001.

In order to investigate pathway components that may act as an escape mechanism while concurrently targeting a downstream kinase that may enable rescue from resistance to EGF-R directed therapies, we propose this prospective, phase II, single-arm, single-agent interventional clinical trial of RAD001 for patients with refractory SCCHN. The primary outcome is activity of RAD001 while secondary outcomes include safety, toxicity and extensive laboratory correlates to be performed on tumor tissues. By carrying out this clinic-translational trial of the novel mTOR inhibitor, RAD001, in patients with refractory SCCHN, we aim to explore mechanisms of activity of and resistance to inhibitors of the EGF-R pathway components while measuring the clinical activity of RAD001.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented squamous cell CA of the head and neck
* Metastatic and/or recurrent head and neck cancer (not eligible for curative intent surgical or radiation therapy)
* Patients must have at least one measurable site of disease according to RECIST criteria that has not been previously irradiated. If the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation
* Performance status 0-2
* Age ≥18 years
* Non-pregnant
* Prior treatment:
* Prior treatment for recurrent or metastatic disease required (at least one): up to but no more than 2 regimens (chemotherapy and/or biologic) allowed.
* Prior induction and concomitant chemoradiotherapy with a curative intent (with or without biologic agents) is allowed
* No other serious medical or psychiatric disease
* Required Lab Values:

Granulocytes ≥ 1,500/µl Platelets ≥ 100,000/µl Bilirubin ≤ 1.5 x ULN INR ≥ 1.3 (or < 3 if on anticoagulation) AST or ALT ≤ 2.5 x ULN (< 5 x ULN in patients with liver metastases) Creatinine ≤ ULN or Creatinine Clearance >= 60 mL/min, if creatinine above ULN

* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* Patients with accessible tumor tissue must agree to a pre-treatment biopsy at screening. If available, original diagnostic tissue may be submitted in place of the pre-treatment biopsy.
* Signed informed consent

Exclusion Criteria:

* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy, etc.)
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study
* Prior treatment with any investigational drug within the preceding 4 weeks
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent, except corticosteroids with a daily dosage equivalent to prednisone ≤ 20 mg. However, patients receiving corticosteroids must have been on a stable dosage regimen for a minimum of 4 weeks prior to the first treatment with RAD001. Topical or inhaled corticosteroids are allowed.
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:
* Symptomatic congestive heart failure of New York heart Association Class III or IV
* unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
* severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air. PFTs as clinically indicated.
* uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
* active (acute or chronic) or uncontrolled severe infections
* liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* A known history of HIV seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active, bleeding diathesis
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes. Hormonal contraceptives are not acceptable as a sole method of contraception. (Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of RAD001)
* Patients who have received prior treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus).
* Patients with a known hypersensitivity to RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus) or to its excipients
* Patients unwilling to or unable to comply with the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-01; Primary Completion 2011-04-26 (Actual); Study Completion 2016-08-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Everolimus 10 mg Daily: Patients with a planned treatment of continuous 28-day cycles of everolimus 10 mg by mouth daily.
Period: Overall Study
Arm/Group | Everolimus 10 mg Daily
Started | 13
Completed | 9
Not Completed | 4
Not completed — Failed screening | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus 10 mg Daily
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 63 [51 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR)
Description: The number of patients with recurrent/refractory SCCHN (head and neck squamous cell carcinoma) treated with single-agent everolimus that, experience a Complete Response (CR) + number of patients that experience a Partial Response (PR ) + number of patients that experience Stable Disease (SD) / total evaluable patients.
Time Frame: Up to 60 months
Population: Patients that completed at least 1 cycle of everolimus treatment.
Measure: Number; unit: percentage of participants
Groups:
- Everolimus 10 mg Daily: Patients that completed at least 1 cycle of everolimus everolimus 10 mg by mouth daily. Response to treatment was evaluated by cross-sectional imaging every 8 weeks or as clinically indicated, starting at the end of cycle 2 and continuing until determination of progressive disease.
Arm/Group | Everolimus 10 mg Daily
Number analyzed (Participants) | 7
percentage of participants | 28

2. Secondary Outcome: Progression Free Survival (PFS)
Time Frame: Up to 60 months
Measure: Median (Full Range); unit: months
Arm/Group | Everolimus 10 mg Daily
Number analyzed (Participants) | 9
months | 1.5 [1.0 to 6.0]

3. Secondary Outcome: Overall Survival (OS)
Time Frame: Up to 60 months
Measure: Median (Full Range); unit: months
Arm/Group | Everolimus 10 mg Daily
Number analyzed (Participants) | 9
months | 4.5 [3.0 to 24.0]

4. Secondary Outcome: Objective Response Rate (ORR)
Description: The number of patients with recurrent/refractory SCCHN (head and neck squamous cell carcinoma) treated with single-agent everolimus that, experience a Complete Response (CR) + number of patients that experience a Partial Response (PR ) / total evaluable patients.
Time Frame: Up to 60 months
Population: Patients that completed at least 1 cycle of everolimus treatment. Response to treatment was evaluated by cross-sectional imaging every 8 weeks or as clinically indicated, starting at the end of cycle 2 and continuing until determination of progressive disease.
Measure: Number; unit: percentage of participants
Arm/Group | Everolimus 10 mg Daily
Number analyzed (Participants) | 7
percentage of participants | 0

ADVERSE EVENTS:
Groups:
- Everolimus 10 mg Daily: Patients with any treatment of everolimus 10 mg by mouth daily.
Arm/Group | Everolimus 10 mg Daily
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 8/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus 10 mg Daily (N=9)
Hemoglobin (Blood and lymphatic system disorders) | 7
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 5
Platelets (Blood and lymphatic system disorders) | 3
Hypotension (Cardiac disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2
Odor (patient odor) (General disorders) | 1
Rigors/chills (General disorders) | 1
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 2
Ulceration (Skin and subcutaneous tissue disorders) | 2
Anorexia (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Dehydration (Gastrointestinal disorders) | 1
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 2
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 5
Mucositis/stomatitis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Salivary gland changes/saliva (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Infection - Other (Specify, __) (Infections and infestations) | 2
Edema: head and neck (Blood and lymphatic system disorders) | 4
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 3
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 5
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 6
Alkaline phosphatase (Metabolism and nutrition disorders) | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 7
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3
Fibrosis-deep connective tissue (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy), Facial (Musculoskeletal and connective tissue disorders) | 1
Trismus (difficulty, restriction or pain when opening mouth) (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Neuropathy: cranial, CN IX Motor-pharynx; Sensory-ear, pharynx, tongue (Nervous system disorders) | 1
Pain - Other (Specify, __) (General disorders) | 3
Pain, Abdomen NOS (General disorders) | 2
Pain, External ear (General disorders) | 1
Pain, Extremity-limb (General disorders) | 2
Pain, Eye (General disorders) | 1
Pain, Face (General disorders) | 2
Pain, Head/headache (General disorders) | 3
Pain, Joint (General disorders) | 1
Pain, Middle ear (General disorders) | 1
Pain, Oral cavity (General disorders) | 2
Pain, Throat/pharynx/larynx (General disorders) | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Obstruction/stenosis of airway, Trachea (Respiratory, thoracic and mediastinal disorders) | 1
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes